CLINICAL TRIAL: NCT02338908
Title: Effectiveness of Dry Needling and Eccentric Exercises in Unspecific Shoulder Pain
Brief Title: Dry Needling and Exercises in Shoulder Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Collaborators: Hospital General Universitario Gregorio Marañon (Other)
Responsible Party: Principal Investigator, César Fernández-de-las-Peñas, Proffesor, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: URJC 31/2140
Record Dates: First submitted 2015-01-11; First posted 2015-01-14 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-03

CONDITIONS: Shoulder Pain
Keywords: dry needling; trigger point; eccentric exercise
MeSH Terms: conditions — Shoulder Pain | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental group (Experimental): Patients will be asked to perform an eccentric loading exercise program for the shoulder musculature, particularly the supraspinatus and infraspinatus muscles, to be performed on an individual basis twice every day. The therapeutic protocol will be applied for 5 weeks. In addition, within the second and fourth sessions, they will receive TrP-DN over active TrPs in the shoulder muscles
  Interventions: Other: exercise program; Other: TrP-DN
- Control group (Active Comparator): Patients will be asked to perform an eccentric loading exercise program for the shoulder musculature, particularly the supraspinatus and infraspinatus muscles, to be performed on an individual basis twice every day. The therapeutic protocol will be applied for 5 weeks.
  Interventions: Other: exercise program

INTERVENTIONS:
Other: exercise program — Patients will be asked to perform an eccentric loading exercise program for the shoulder musculature, particularly the supraspinatus and infraspinatus muscles, to be performed on an individual basis twice every day. The therapeutic protocol will be applied for 5 weeks.
Other: TrP-DN — In addition, within the second and fourth sessions, they will receive TrP-DN over active TrPs in the shoulder muscles
  Arms: Experimental group

SUMMARY:
Shoulder pain is highly prevalent in the society. The role of muscle tissues in this pathology has received increasing interest. Some studies have proposed the role of myofascial trigger points in this population. The purpose of the current clinical trial is to compare the effects of physiotherapy treatment consisting of an eccentric exercise protocol versus the same physical therapy program plus the addition of trigger point dry needling (TrP-DN) on pain and function in patients suffering from unspecific shoulder pain.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral non-traumatic shoulder pain
* Shoulder pain from at least 3 months
* Shoulder pain of more than 4 points on a NPRS

Exclusion Criteria:

* bilateral shoulder symptoms
* younger than 18 or older than 65 years
* history of shoulder fractures or dislocation
* cervical radiculopathy
* previous interventions with steroid injections
* fibromyalgia syndrome
* previous history of shoulder or neck surgery
* any type of intervention for the neck-shoulder area during the previous year

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Changes in disability between baseline and follow-up periods | Baseline, one week after the last intervention and 3, 6 and 12 months after the intervention
  The Disabilities of the Arm, Shoulder and Hand (DASH) will be used to determine the disability induced by shoulder pain

SECONDARY OUTCOMES:
Changes in shoulder pain between baseline and follow-up periods | Baseline, one week after the last intervention and 3, 6 and 12 months after the intervention
  A 10-point Numerical Pain Rating Scale (NPRS; 0: no pain, 10: maximum pain) will be used to assess the patients' current level of shoulder pain and the worst level of pain experienced in the preceding week in the shoulder area.

CONTACTS AND LOCATIONS:
Overall Officials: César Fernández-de-las-Peñas, PT, PhD, Principal Investigator — Universidad Rey Juan Carlos
Locations (1):
- César Fernández-de-las-Peñas, Alcorcón, Madrid, Spain

REFERENCES:
- [Derived] Arias-Buria JL, Fernandez-de-Las-Penas C, Palacios-Cena M, Koppenhaver SL, Salom-Moreno J. Exercises and Dry Needling for Subacromial Pain Syndrome: A Randomized Parallel-Group Trial. J Pain. 2017 Jan;18(1):11-18. doi: 10.1016/j.jpain.2016.08.013. Epub 2016 Oct 5. PMID 27720812